CLINICAL TRIAL: NCT01559337
Title: Nerve Transfer for Finger Sensory Reconstruction With Dorsal Branch of the Digital Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEN-19750471
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Sensory Restoration of the Reconstructed Finger Pulps; Cold Intolerance of the Reconstructed Finger; Pain of the Reconstructed Finger
Keywords: defect; dorsal branch of the proper digital nerve; proper digital nerve; nerve transfer; finger sensory reconstruction
MeSH Terms: interventions — Nerve Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nerve repair (Other): the dorsal branch of the proper digital nerve was used as a pedicle nerve for reconstructing PDN defects
  Interventions: Procedure: Nerve transfer

INTERVENTIONS:
Procedure: Nerve transfer — the dorsal branch was used as a pedicle nerve for reconstructing PDN defects
  Other Names: Local pedicle nerve transfer

SUMMARY:
A proper digital nerve (PDN) defect causes partial or complete sensory loss of the finger pulp, which results in functional disability.The dorsal branch of the PDN can be transferred for reconstruction of such nerve defects.In this study, the investigators modified the Lesavoy et al' technique and evaluated the efficacy of dorsal sensory branch transfer for PDN defects. For comparison, the investigators collected a consecutive series of 32 patients with finger PDN defects treated using a traditional sural nerve graft from February 2005 to October 2008.

ELIGIBILITY:
Inclusion Criteria:

1. Finger PDN defects proximal to the proximal interphalangeal joint
2. Single or two PDN defects
3. PDN defects longer than 1 cm.

Exclusion Criteria:

1. PDN defects less than 1 cm
2. Concomitant injuries to the multiple dorsal sensory branches that preclude their use as nerve donor sites
3. Thumb PDN defects.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination (2PD) test | 26 months
  At final follow-up, we measured the sensibility of the pulps and the donor sites using the static 2-point discrimination (2PD) test. The test points were at the center of the radial or ulnar portion of the pulp and the donor sites separately. Each area was tested 3 times with a Dellon-Mackinnon discriminator. Two out of 3 correct answers were considered proof of perception before proceeding to another lower value.

SECONDARY OUTCOMES:
self-administered Cold Intolerance Severity Score (CISS) questionnaire | 26 months
  The maximum score was 100 and was grouped into 4 ranges (0-25, 26-50, 51-75, and 76-100), corresponding to mild, moderate, severe, and extreme severity, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Peifu Tang, MD., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Ethetic Committee of Tangshan, Tangshan, Hebei, China